CLINICAL TRIAL: NCT02016235
Title: Role Of Phosphorus And FGF 23 In Patients With Dent Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-004774
Record Dates: First submitted 2013-12-06; First posted 2013-12-19 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Dent Disease
Keywords: Dent; Dents; Dent Disease; Phosphorus Supplements; FGF 23
MeSH Terms: conditions — Dent Disease | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dent Disease Intervention (Experimental): Dent Disease subjects will receive 2 week supplementation with phosphorus
  Interventions: Drug: Phosphorus Supplement
- Kidney Stone subjects (Experimental): Kidney stone with or without phosphate leak subjects will receive 2 week supplementation with phosphorus
  Interventions: Drug: Phosphorus Supplement
- Dent Disease Observation (Placebo Comparator): Dent disease subjects will not get phosphorus
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Phosphorus Supplement — 250 mg po qid
  Other Names: K-phos neutral
  Arms: Dent Disease Intervention; Kidney Stone subjects
Other: Observation — Baseline blood and urine measurements only
  Arms: Dent Disease Observation

SUMMARY:
Patients with Dent disease have suppressed levels of FGF 23 which contributes to hypercalciuria, kidney stones, nephrocalcinosis and renal failure. Supplementation with phosphorus may reduce hypercalciuria.

ELIGIBILITY:
Inclusion Criteria:

Patients will be recruited from those in the RKSC Dent Registry

1. Diagnostic criteria for Dent disease Observational arm include:

   1. <18 years old
   2. LMWP (at least 5 times above the upper limit of normal) and at least 1 of the following criteria: 1. Hypercalciuria, 2. Kidney stones, 3. Nephrocalcinosis, 4. Hypophosphatemia, 5. Renal phosphate leak, 6. Aminoaciduria, 7. Glucosuria without diabetes mellitus, 8. Hematuria, 9. Renal insufficiency, 10. Family history with x-linked inheritance or
   3. 1 of the above criteria (1-9) and confirmed genetic mutation of CLCN5 or OCRL1.
2. Diagnostic criteria for Dent disease Intervention arm include:

   1. >18 years old
   2. LMWP (at least 5 times above the upper limit of normal) and at least 1 of the following criteria: 1. Hypercalciuria, 2. Kidney stones, 3. Nephrocalcinosis, 4. Hypophosphatemia, 5. Renal phosphate leak, 6. Aminoaciduria, 7. Glucosuria without diabetes mellitus, 8. Hematuria, 9. Renal insufficiency, 10. Family history with x-linked inheritance or
   3. 1 of the above criteria (1-9) and confirmed genetic mutation of CLCN5 or OCRL1.
3. Idiopathic calcium nephrolithiasis with renal phosphate leak

   1. Male patients > 18 years old
   2. History of symptomatic calcium oxalate or calcium phosphate stone, hypercalciuria (>250 mg/24 hrs), renal phosphate leak (TMP/GFR <2.07 mg/dl)
4. Idiopathic calcium nephrolithiasis without renal phosphate leak

   1. Male patients > 18 years old
   2. History of symptomatic calcium oxalate or calcium phosphate stone, hypercalciuria (>250 mg/24 hrs), renal phosphate leak (TMP/GFR <2.07 mg/dl)

Exclusion Criteria:

1. Exclusion for Dent disease include: primary or secondary hyperparathyroidism, hyperthyroidism, chronic diarrhea states; intake of thiazide diuretics, glucocorticoids, or estrogens within one month of the study.
2. Exclusion criteria for calcium stone formers include: primary or secondary hyperparathyroidism, hyperthyroidism, estimated GFR <40 ml/mn/1.73m2, chronic diarrhea states; intake of thiazide diuretics, glucocorticoids, or estrogens within one month of the study.
3. Exclusion criteria include history of symptomatic or asymptomatic kidney stone disease; primary or secondary hyperparathyroidism; estimated GFR <40 ml/min/1.73m2, chronic diarrhea states; intake of thiazide diuretics, glucocorticoids, or estrogens within one month of the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dent Disease Intervention | Kidney Stone Subjects | Dent Disease Observation
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dent Disease Intervention | Kidney Stone Subjects | Dent Disease Observation | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (12.0) | 55.3 (14.6) | 10.2 (1.3) | 30.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Total Protein
Description: Urine protein tests detect and/or measure protein being released into the urine. Normal urine protein elimination is less than 150 mg/day
Time Frame: baseline, day 7
Population: Data were not collected for the Disease Dent Observation Group
Measure: Mean (Standard Deviation); unit: mg/day
Groups:
- Dent Disease Observation: Dent disease subjects will not get phosphorus
  Observation: Baseline blood and urine measurements only. Day 7 Urine total protein not obtained
Arm/Group | Dent Disease Intervention | Kidney Stone Subjects | Dent Disease Observation
Number analyzed (Participants) | 10 | 10 | 0
mg/day | 1681 (979) | 59 (38) |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a period of 7 days for each subjects
Arm/Group | Dent Disease Intervention | Kidney Stone Subjects | Dent Disease Observation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02016235/Prot_SAP_000.pdf